CLINICAL TRIAL: NCT01736644
Title: A Prospective Randomized Control Trial to Compare the Aquamantys System With Standard Electrocautery in Reducing Blood Loss in Primary Total Knee Arthroplasty
Brief Title: Bipolar Sealer Aquamantys Use in Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TD-07709
Record Dates: First submitted 2012-11-20; First posted 2012-11-29 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis; Arthritis; Surgery; Infection; Inflammation; Disability; Hemorrhage
Keywords: blood loss; bipolar sealer; aquamantys; total knee replacement; primary total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis; Infections; Inflammation; Hemorrhage | interventions — Electrocoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrocautery (Placebo Comparator): Use of electrocautery in tourniquet and without tourniquet total knee replacement surgery.
  Interventions: Device: Electrocautery
- Bipolar Sealer Aquamantys (Active Comparator): Use of bipolar sealer Aquamantys in tourniquet and tourniquetless total knee replacement surgical procedures.
  Interventions: Device: Bipolar sealer Aquamantys

INTERVENTIONS:
Device: Electrocautery — Use of electrocautery in tourniquet and tourniquetless total knee replacement surgery
  Arms: Electrocautery
Device: Bipolar sealer Aquamantys — Aquamantys use in tourniquet and tourniquetless total knee replacement.
  Other Names: Aquamantys; AQM; Bipolar sealer
  Arms: Bipolar Sealer Aquamantys

SUMMARY:
This study will compare the clinical outcomes for patients undergoing a total knee replacement using a bipolar sealer, the Aquamantys® System, as compared to standard electrocautery. Total blood loss during the hospital stay and knee mobility and discharge factors will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 years of age
* Patient has failed conservative therapy of osteoarthritis of the knee and has been listed to undergo primary TKA
* Patient is willing and able to provide written informed consent.
* Pre-assessment Haemoglobin ≥ 11.0g/dl
* Patient is suitable to receive spinal anaesthesia with no peripheral nerve blocks
* Patients willing to undergo blood transfusion

Exclusion Criteria:

* Patients that are listed for unicondylar or revision TKA
* Patients who are being converted from a previous high tibial osteotomy and a previous unicondylar knee arthroplasty
* Fixed motor deficit thus affecting functional assessment of the knee
* Patients presenting with a non-osteoarthritis degenerative knee diagnosis
* Patients presenting with known contralateral knee osteoarthritis requiring simultaneous bilateral TKA
* Patients presenting with a history of previous knee infection
* Patients presenting with a pre-operative knee range of motion < 85°
* Knee deformity greater than 20 degrees varus or valgus
* Patients presenting with a history of bleeding disorders and/or are on chronic blood anticoagulation therapy
* Patients with significantly impaired renal function (defined by EGFR >30)
* Patients with allergy or sensitivity to non-steroidal anti-inflammatory drugs, ropivacaine, ketoprofen or adrenaline
* Patients presenting with an internal cardiac defibrillator
* Women who are pregnant
* Evidence of active (systemic or local) infection at time of surgery
* Patients who have habitual opioid use
* Patients who have a psychiatric or mental illness which could impair the consent process or ability to complete patient-report questionnaires
* Morbid obesity [BMI > 40]
* Patients who are unwilling to undergo blood transfusion, if necessary
* Patients who are receiving any implant used in conjunction with a customised-cutting block system
* Any patient who cannot or will not provide written informed consent for participation in the study
* Those whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-10-27 (Actual); Study Completion 2013-10-27 (Actual)

PRIMARY OUTCOMES:
Blood Loss | upto to 72 hrs after surgery
  The primary outcome will be total blood loss throughout the hospital stay.

SECONDARY OUTCOMES:
Rehabilitation | 6-weeks
  Discharge criteria evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Field, Md, PhD, FRCS, Principal Investigator — SWLEOC
Locations (2):
- United Kingdom (2):
  - South West London Elective Orthopaedic Center, Epsom, Surrey
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Background] Marulanda GA, Krebs VE, Bierbaum BE, Goldberg VM, Ries M, Ulrich SD, Seyler TM, Mont MA. Hemostasis using a bipolar sealer in primary unilateral total knee arthroplasty. Am J Orthop (Belle Mead NJ). 2009 Dec;38(12):E179-83. PMID 20145794
- [Background] Marulanda GA, Ragland PS, Seyler TM, Mont MA. Reductions in blood loss with use of a bipolar sealer for hemostasis in primary total knee arthroplasty. Surg Technol Int. 2005;14:281-6. PMID 16525984
- [Background] Pfeiffer M, Brautigam H, Draws D, Sigg A. A new bipolar blood sealing system embedded in perioperative strategies vs. a conventional regimen for total knee arthroplasty: results of a matched-pair study. Ger Med Sci. 2005 Dec 13;3:Doc10. PMID 19675727